CLINICAL TRIAL: NCT01286766
Title: A Randomized Phase II Trial of Neoadjuvant Combination Chemotherapy of DCS (Cisplatin + Docetaxel + S-1) and DCF (Docetaxel + Cisplatin + 5-FU) in Patients With Locally Advanced Gastric Adenocarcinoma
Brief Title: Neoadjuvant Combination Chemotherapy of DCS and DCF in Patients With Locally Advanced Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2009-0332
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer
Keywords: unresectable; locally advanced
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cycloserine; Docetaxel; Cisplatin; titanium silicide; Pentostatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCS (Active Comparator): DCS: docetaxel with cisplatin with TS-1
  Interventions: Drug: DCS (docetaxel with cisplatin with TS-1)
- DCF (Active Comparator): DCF : docetaxel with cisplatin with 5-FU
  Interventions: Drug: DCF (docetaxel with cisplatin with 5-FU)

INTERVENTIONS:
Drug: DCS (docetaxel with cisplatin with TS-1) — 1. S-1: 70 mg/m2 #2 bid PO, D1-14
  2. Docetaxel 30 mg/m2 IVF (for 1 hr) D1 and D8
  3. Cisplatin 30 mg/m2 IVF (for 2 hrs, without hydration) D1 and D8, repeated by 3 weeks.
  Other Names: Taxotere; CDDP; TS-1
  Arms: DCS
Drug: DCF (docetaxel with cisplatin with 5-FU) — 1. 5-FU: 1,000 mg/m2 CI, D1-3
  2. Docetaxel 60 mg/m2 IVF (for 1 hr) D1 followed by
  3. Cisplatin 60 mg/m2 IVF (for 2 hrs, with hydration) D1, repeated by 3 weeks.
     * Intercycle or intracycle dose modification is indicated if ≥G3 hematologic toxicity (except anemia) or ≥G3 non-hematologic toxicity (except alopecia)
     * treatment is repeated until 4 cycles
  Other Names: 5-FU; Taxotere; CDDP
  Arms: DCF

SUMMARY:
Number of patients planned The study adopted two parallel phase II studies, with the same P1 and P0 in each arm, suggested by Logan. The investigators hypothesized a target ORR of interest, P1=50, and a lower ORR, P0=25 with the treatment of DCS and DCF, respectively. Under the assumption of α-error=0.05 and β-error= 0.2, using sample size tables of A'Hern, 26 patients were required per arm to achieve the desired statistical power. Finally, taking a 20% drop-out rate into consideration, the overall number of enrolled patients was 62.

DETAILED DESCRIPTION:
Treatment scheme

* Screening period: D-21 to D1 (treatment day)
* Preoperative screening includes EUS, laparoscopy (optional), EGD and abd-pelvic CT scan.
* Preoperative clinical staging is based on the guideline of Japanese Gastric Cancer Association (JGCA, 1998)
* Tumor response is assessed every 2 cycles (6 weeks)
* Treatment is repeated until,.

  * 4 cycles
  * progressive disease
  * unacceptable toxicity
  * patient's withdrawal
* Gastric surgery should be performed within 4~6 weeks of the last dose of chemotherapy
* Gastric surgery is for curative aim and should include ≥ D2 LN dissection.
* Patients who received R0 resection should receive at least 4-cycled adjuvant chemotherapy with 5-FU and cisplatin.
* Palliative chemotherapy should be indicated for inoperable progressive disease or who failed curative resection. 5-FU and oxaliplatin combination is recommended as first-line therapy.
* Follow up for survival is repeated every 3 months for 2 years

Study period Patient enroll period for 12 months., and follow-up duration for further 12 months., resulting total study period of 24 months

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed gastric adenocarcinoma
* Age 18 to 70 years old
* ECOG performance Status 0~1
* Preoperative clinical staging by Japanese Gastric Cancer Association (JGCA): cT3N2 (IIIB), cT4N0-3 (IIIA~IV), M0, P0, H0, CY0
* No pretreatment (radiotherapy or chemotherapy) for gastric cancer
* Adequate organ function

  * Hb ≥ 9.0 g/dL
  * WBC ≥ 4,000/µL
  * ANC ≥ 2,000/µL (*ANC = Neutrophil segs ＋ Neutrophil bands)
  * Platelet ≥ 100 × 103/ µL
  * Total bilirubin: ≤ 1.5 × UNL
  * CCr ≥ 60 ml/min (by laboratory or Cockcroft-Gault Formula)
  * AST/ALT, ALP: ≤ 2.5 × UNL
* Written informed consent

Exclusion Criteria:

* Distant metastasis on diagnosis
* cT1-2
* Cancer of gastroesophageal junction (GEJ)
* Poor oral intake or absorption deficiency syndrome
* Gastric outlet obstruction, perforation or bleeding
* Medically uncontrollable chronic illness or infection
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* History of clinically significant cardiac disease
* Past or concurrent history of neoplasm last < 5 year other than gastric cancer
* Prior gastrectomized patients
* Concomitant administration of any other experimental drug under investigation
* Peripheral neuropathy ≥ NCI-CTC grade 2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
RECIST(Response Evaluation Criteria in Solid Tumors) | written in the description part below
  * safety : every cycle adverse event/serious adversr event evaluation from NCI-CTC(version 3.0)
  * efficacy : tumor response is assessed every 2 cycles (6weeks) -> tumor response assessment(RECIST<Response Evaluation Criteria in Solid Tumor> 1.0 version use)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea